CLINICAL TRIAL: NCT01068769
Title: A Multi-center Phase II Study Evaluating the Efficacy and Safety of Regorafenib in Patients With Metastatic and/or Unresectable Gastrointestinal Stromal Tumor (GIST), Resistent or Intolerant to at Least Imatinib and Sunitinib
Brief Title: Regorafenib in Patients With Metastatic and/or Unresectable Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzanne George, MD (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Fox Chase Cancer Center (Other); Oregon Health and Science University (Other); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Suzanne George, MD, Clinical Director Center for Sarcoma and Bone Oncology, Dana-Farber/Brigham and Women's Cancer Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-400
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: regorafenib; GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib (Experimental): Regorafenib adminstered orally, 160 mg per day on days 1 through 21 of a 28 day cycle
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib — Taken orally, once a day in the morning for 3 weeks followed by a one week rest period
  Other Names: Stivarga

SUMMARY:
The purpose of this research study is to determine the safety and activity of regorafenib in participants with advanced gastrointestinal stromal tumor (GIST) if the standard approved therapies, imatinib and sunitinib, have failed to control the disease. Regorafenib is a drug that blocks abnormally active signaling enzymes called "tyrosine kinases" which are important to the growth of GIST. This "tyrosine kinase inhibition" is similar to the way that both imatinib and sunitinib work; however, regorafenib blocks certain additional signaling pathways that are not blocked by imatinib or sunitinib. Regorafenib has been not been tested in GIST participants before this research study.

DETAILED DESCRIPTION:
* In this research study, each planned "cycle" of the study lasts 4 weeks. In the first cycle, participants will come to the clinic on Days 1, 15 and 16. For cycles 2 through 4, they will come to the clinic on Days 1 and 15 of each cycle. For cycle 5 and beyond, they will come to the clinic on Day 1 of each cycle. Repeat tumor imaging will be performed at the end of every 2 cycles during study drug administration (e.g. end of cycles 2, 4, 6, etc.)
* During each cycle, participants will take regorafenib by mouth, once a day in the morning, for 3 weeks followed by one week during which you do not take regorafenib (the "rest period").
* FDG-PET/CT (Positron Emission Tomography) scans are required as part of this study to monitor effects of the study drug on the participant's GIST. The first scan will take place before the first dose of study drug. If the first scan shows that the "tracer sugar" collection is increased in the participant's GIST, they will have up to 5 additional scans performed at different time points throughout their participation in this research study.
* Participants may continue to participate in this research study for as long as they do not have serious side effects or their disease does not get worse.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of study entry
* Histologically confirmed metastatic and/or unresectable GIST with prior failure of both conventional tyrosine kinase inhibitors, imatinib and sunitinib.
* Measurable disease per RECIST 1.1. A lesion in a previously irradiated area is eligible to be considered as measurable disease as long as there is objective evidence of progression of the lesion.
* ECOG Performance Status 0 or 1
* Adequate organ and marrow function as outlined in the protocol
* Fully recovered from the acute effects of prior cancer therapy before initiation of study drug
* Patients must be suitable for oral drug administration
* Willingness to use effective means of birth control throughout the duration of clinical study and for at least 3 months after completion of study drug
* Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of study drug administration

Exclusion Criteria:

* Use of any unapproved tyrosine kinase inhibitors or investigational agents within 2 weeks or 6 half-lives of the agent, whichever is shorter, prior to receiving study drug
* Participants who have had radiotherapy within 4 weeks prior to study entry
* Major surgery, or significant traumatic injury within 4 weeks prior to study entry
* Presence of symptomatic or uncontrolled brain or central nervous system metastases
* Prior exposure to sorafenib
* Prior exposure to regorafenib
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Individuals with a history of a different malignancy, other than cervical cancer in situ, basal cell or squamous cell carcinoma of the skin, are ineligible, except if they have been disease-free for at least 5 years, and are deemed by the investigator to be at low risk for recurrence of that malignancy or other primary malignancy is neither currently clinically significant nor requiring active intervention
* Clinically significant cardiac arrhythmias and/or patients who require anti-arrhythmic therapy (excluding beta blockers or digoxin)
* History of clinically significant cardiac disease or congestive heart failure > NYHA class 2. Patients must not have unstable angina or new-onset angina within the last 3 months or myocardial infarction within the past 6 months
* Hypertension as defined by systolic blood pressure 140-159 mmHg or diastolic blood pressure 90-99 mmHg; recurrent or persistent or symptomatic increase by > 20 mmHg (diastolic) or to systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg if previously within normal limits, despite optimal medical management
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before start of study medication
* Ongoing infection of Grade 3 or higher
* Patients with evidence of, or history of, bleeding diathesis. Any major hemorrhage or bleeding event of Grade 3 or higher within 4 weeks of start of study medication
* Non-healing wound, ulcer or bone fracture
* Renal failure requiring hemo-or peritoneal dialysis
* Dehydration of Grade 2 or greater
* Persistent proteinuria Grade 3 or higher
* Known history of HIV infection or chronic hepatitis B or C
* Uncontrolled intercurrent illness
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne George, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Oregon Health Sciences University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Ben-Ami E, Barysauskas CM, von Mehren M, Heinrich MC, Corless CL, Butrynski JE, Morgan JA, Wagner AJ, Choy E, Yap JT, Van den Abbeele AD, Solomon SM, Fletcher JA, Demetri GD, George S. Long-term follow-up results of the multicenter phase II trial of regorafenib in patients with metastatic and/or unresectable GI stromal tumor after failure of standard tyrosine kinase inhibitor therapy. Ann Oncol. 2016 Sep;27(9):1794-9. doi: 10.1093/annonc/mdw228. Epub 2016 Jul 1. PMID 27371698

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at three sites between February and December, 2010.
Period: Overall Study
Arm/Group | Regorafenib
Started | 34
Completed | 33
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients were included in the baseline analysis population
Arm/Group | Regorafenib
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 56 [25 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit as Defined by the Composite of Complete Response, Partial Response and Stable Disease Lasting 16 Weeks or More Per RECIST 1.1 as a Measure of Disease Control
Description: The composite of complete response, partial response, and stable disease lasting 16 weeks or more per RECIST 1.1 as a measure of disease control. This is for target lesions. Complete response is disappearance of all target lesions and partial response is >+30% decrease in the sum of the longest diameter of target lesions. Stable disease is neither shrinkage by greater than or equal to 30% of the sum of the longest diameter of target lesions or the increase of lesions by greater than or equal to 20% of the sum of the longest diameter of target lesions. Progressive disease is considered an increase of the sum of the longest diameter of target lesions by greater than or equal to 20%.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 33
percentage of participants | 75 [61 to 91]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the duration of time from start of study drug administration to time of objective disease progression or death due to any cause, whichever comes first. Progression is evaluated every 8 weeks using Response Criteria for Solid Tumors (RECIST) 1.1. Objective disease progression is defined as a 20% increase in the sum of the longest diameter of target lesion(s).
Time Frame: From date of enrollment until date of first documented progression or date of death from any cause, whichever came first
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib
Number analyzed (Participants) | 33
months | 10.0 [8.3 to 14.9]

ADVERSE EVENTS:
Arm/Group | Regorafenib
Serious Adverse Events (participants affected / at risk) | 31/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regorafenib (N=33)
Acute coronary syndrome (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Colitis (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 2
Blood bilirubin increased (Investigations) | 1
CD4 lymphocytes decreased (Investigations) | 1
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Serum amylase increased (Investigations) | 1
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Insomnia (Psychiatric disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 13
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regorafenib (N=33)
Leukocytosis (Blood and lymphatic system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 9
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 5
Eye disorders - Other, specify (Eye disorders) | 3
Bloating (Gastrointestinal disorders) | 2
Oral dysesthesia (Gastrointestinal disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 8
Colitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 23
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 8
Flatulence (Gastrointestinal disorders) | 7
Mucositis oral (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 13
Oral hemorrhage (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 3
Stomach pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 9
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 19
Chills (General disorders) | 2
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 26
Pain (General disorders) | 2
Mucosal infection (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 4
Creatinine increased (Investigations) | 2
Lipase increased (Investigations) | 6
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 4
Serum amylase increased (Investigations) | 3
Weight loss (Investigations) | 7
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 15
Urinary frequency (Renal and urinary disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 18
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 18
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Scalp pain (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4
Flushing (Vascular disorders) | 2
Hot flashes (Vascular disorders) | 3
Hypertension (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No